CLINICAL TRIAL: NCT01663688
Title: Normative Data Collection Study of the Nidek Optical Coherence Tomography RS-3000 for the Measurements of Retinal and RNFL Thickness and Optic Disc Analysis
Brief Title: Data Collection Study of the Nidek Optical Coherence Tomography RS-3000 for 3D Measurements of the Eye
Status: Completed | Type: Observational
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: OCT RS-3000
Record Dates: First submitted 2012-07-12; First posted 2012-08-13 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Ocular Physiology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normative Data Collection

SUMMARY:
The purpose of this clinical study is to collect and evaluate the data from eye scans using an investigational three-dimensional eye imaging photography device called the Nidek Optical Coherence Tomography (OCT) RS-3000. OCT stands for Optical Coherence Tomography, a technique that uses invisible wavelengths of light to make detailed images of the tissues at the back of the eye. These images provide information that physicians may use to help diagnose eye conditions and/or to monitor changes in the eye during treatment.

DETAILED DESCRIPTION:
This is a prospective, open-labeled, multi-center clinical study. After qualifying examination of a subject, 3D retinal measurement in the proximity of the optic disc and the macula are carried out for eligible subjects with normal eyes using an investigational three-dimensional eye imaging photography device called the Nidek Optical Coherence Tomography (OCT) RS-3000. The primary objective of this clinical study is to develop age-specific normal ranges for the thickness of the retina and retinal nerve fiber layer (RNFL) etc. using the Nidek Optical Coherence Tomography (OCT) RS-3000 with normative database. The secondary objective is to evaluate any adverse events found during the clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Normal and healthy male and female subjects at least 20 years of age.

Exclusion Criteria

* Subjects who have extensive or debilitating systemic diseases.
* Subjects who have significant ocular disease.
* Subjects who are extremely far sighted or extremely near sighted.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal subject eyes
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Development of age-specific normal ranges for the thickness of the retina and retinal nerve fiber layer (RNFL) and Optic Disc Analysis | Subjects will be followed for the duration of the procedure, up to one day.
  The primary objective of this clinical study is to develop age-specific normal ranges for the thickness of the retina and retinal nerve fiber layer (RNFL)and Optic Disc Analysis.

SECONDARY OUTCOMES:
Evaluation of adverse events found during the clinical study | Subjects will be followed for the duration of the procedure, up to one day.
  The secondary objective is to evaluate any adverse events found during the clinical study.

CONTACTS AND LOCATIONS:
Overall Officials: Robert N Weinreb, MD, Principal Investigator — Hamilton Glaucoma Center, UC San Diego
Locations (3):
- United States (3):
  - UC San Diego, Hamilton Glaucoma Center, Department of Ophthalmology, La Jolla, California
  - USC Eye Institute, Keck Medical Center of USC, Los Angeles, California
  - UC Davis, Medical Center, Department of Ophthalmology & Vision Science, Sacramento, California